CLINICAL TRIAL: NCT01423370
Title: Multi-center, Randomized, Double-blind, Placebo/Active-controlled, Phase II Clinical Trial to Assess the Safety and Efficacy of YHD1023 in Patients With Erectile Dysfunction
Brief Title: Safety and Efficacy of YHD1023 in Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YHD1023-201
Record Dates: First submitted 2011-08-24; First posted 2011-08-25 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2013-05

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; YHD1023; YCD190; Cialis; Yuhan
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Experimental)
  Interventions: Drug: YHD1023
- Group B (Experimental)
  Interventions: Drug: YHD1023
- Group C (Experimental)
  Interventions: Drug: YHD1023
- Group D (Active Comparator)
  Interventions: Drug: Cialis
- Group E (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YHD1023 — 5g oral once daily
  Arms: Group A
Drug: YHD1023 — 5g oral twice a day
  Arms: Group B
Drug: YHD1023 — 10g oral once daily
  Arms: Group C
Drug: Cialis — 5mg oral once daily
  Arms: Group D
Drug: Placebo — Oral
  Arms: Group E

SUMMARY:
The objective of this study is to assess the safety and efficacy of oral YHD1023 5g or 10g on erectile dysfunction to investigate the optimal recommended dosage. Study period is 12 weeks including 4weeks of follow-up period without treatment. Study patients will fill in the international index of erectile function questionnaire and life satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers of aged 20 years and older with history of organic erectile dysfunction of at least 6 months duration
* Anticipate having the same adult female sexual partner, who have no possibility of being pregnant or breast-feeding and take steps to prevent conception during the study
* The patient or legally authorized representative must sign a written informed consent, prior to the any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the purpose, contents, and characteristic of the drug
* Have Erectile Function(EF) domain score 25 and under as the result of the International Index of Erectile Function(IIEF)
* Agree to make at least 4 sexual intercourse attempts on 4 separate days with the female sexual study party during the 4-week run-in period without medication and at least 50% of attempts during this period had been unsuccessful due to insufficient erection or unable to sustain penile rigidity until ejaculation

Exclusion Criteria:

* Have history of stroke, myocardial infarction, or Coronary Artery Bypass Graft surgery within the last 6 months
* Have history of cardiac failure, unstable angina, or life-threatening arrhythmia within the last 6 months
* Shown tachyarrhythmia, heart rate over 100 times/min(e.g. arterial fibrillation, flutter)
* Presence of hypotension as evidenced by SBP/DBP < 90/50mmHg or uncontrollable hypertension as evidenced by SBP/DBP > 170/100mmHg
* Presence of diagnosed diabetes(HbA1C > 12%)
* Have history of symptomatic postural hypotension within the last 6 months
* Have history of spinal cord injury, radical prostatectomy, or pelvic surgery
* Presence of penile anatomical deformities (e.g. severe penile fibrosis or Peyronie's disease)
* Presence of hypogonadism(serum total testosterone under the reference lowest limit)
* Presence of hepatic impairment(AST or ALT > 3 times of normal upper limit) or renal impairment(serum creatinine ≥ 2.5mg/dl)
* Have history of severe gastrointestinal hemorrhage within the last 1 year
* Have history of hematodyscrasia predisposing to priapism(e.g. sickle cell disease, multiple myeloma, or leukemia) or bleeding disorder
* Subject who is judged to be ineligible according to their physical checkup(medical history, physical examination, ECG, laboratory values and etc.) within 56 days prior to the first administration
* Concomitant use of one or more of nitrates/nitric oxide(NO) donor(e.g. nitroglycerine, isosorbid, mononitrate, isosorbid dinitrate, amylnitrate/nitrite, sodium nitroprusside), Trazodone, cancer chemotherapy, anticoagulants, androgens, or anti-androgens
* Use of any PDE-5 inhibitor(e.g. Viagra, Levitra, Cialis, Yaila, or Zydena), vasodilator self-injection, or other treatments for erectile dysfunction within the last 2 weeks prior to the study
* Participated in any other clinical trials within 30 days prior to the first administration
* Have history of primary hypoactive sexual desire
* Subject who is judged to be ineligible by principal investigator or sub-investigator due to mental disorder or continuous drug abuse

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the International Index of Erectile Function(IIEF) - Erectile Function(EF) domain score at week 8 | Baseline, Week 8

SECONDARY OUTCOMES:
Percentage of Improved patients from baseline in Question 3 & Question 4 of the International Index of Erectile Function(IIEF) at week 8 | Baseline, Week 8
  *Improved: Score increased 1 or more compared to the baseline score
  Question 3: How many times were you able to insert your penis into your partner's vagina? Scores range from 0(did not have sexual intercourse) to 5(always or most times).
  Question 4: How many times did your erection last long enough for you to complete intercourse? Scores range from 0(did not have sexual intercourse) to 5(always or most times).
Mean change from baseline in other Question of International Index of Erectile Function(IIEF) domain at week 8 | Baseline, Week 8
Percentage of Improved patients from baseline in Question 2 & Question 3 of Sexual Encounter Profile(SEP) at week 8 | Baseline, Week 8
  *Improved: Response change from "No" at baseline to "Yes" at week 8
  Question 2: Were you able to insert your penis into your partner's vagina?
  Question 3: Did your erection last long enough for you to complete intercourse with ejaculation?
Percentage of Improved patients from baseline in Global Assessment Question(GAQ) at week 8 | Week 8
  *Improved: Yes response at week 8
  GAQ: Did the 4 week treatment improve you ability to achieve and maintain your erection?
Mean change in Life Satisfaction score | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Cheol Park, MD, PhD., Principal Investigator — Busan National University Hospital
Locations (1):
- Yuhan Corporation, Seoul, South Korea